CLINICAL TRIAL: NCT00854477
Title: A Pharmacokinetic Study of Adjuvant Capecitabine in Patients Who Have Undergone Proximal Pancreatico-duodenectomy for Resection of Pancreatic Adenocarcinoma
Brief Title: Pharmacokinetic Study of Adjuvant Capecitabine After Resection of Pancreatic Adenocarcinoma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Duncan Jodrell, Professor Duncan Jodrell, Cambridge University Hospitals NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CAP001; PDDG/CAP001
Record Dates: First submitted 2009-02-27; First posted 2009-03-03 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: capecitabine; Post whipples; pancreatico-duodenectomy; pancreatic adenocarcinoma; pharmacokinetic
MeSH Terms: interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: capecitabine — film-coated tablet 1250 mg/m2 twice daily for 14 days every 3 weeks. Number of cycles: 8 cycles unless there is evidence of disease progression, or unacceptable toxicity
  Other Names: Xeloda

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (PK) of adjuvant capecitabine in patients who have undergone proximal pancreatico-duodenectomy.

DETAILED DESCRIPTION:
Primary Objective:

* To establish the pharmacokinetics (PK) of capecitabine in patients who have undergone proximal pancreatico-duodenectomy.

Secondary objectives:

* To establish the toxicity profile of capecitabine in these patients and to identify any dose limiting toxicities (DLT).
* To ensure equivalent capecitabine exposure when compared to previous studies using patients who have not undergone such surgery.

This is a clinical trial to evaluate the pharmacokinetics (PK) of adjuvant capecitabine in patients who have undergone proximal pancreatico-duodenectomy. The study also aims to establish the toxicity profile of capecitabine in these patients, to identify any dose limiting toxicities (DLT), and to ensure equivalent capecitabine exposure when compared to previous studies using patients who have not undergone such surgery. Screening tests will consist of demographic details, complete medical history, physical exam, vital signs, tumour serum markers, haematology and biochemistry tests. There will also be an ECG, faecal elastase measurement and a serum or urine pregnancy test (for women of childbearing potential). Haematology and Biochemistry (including CA19.9) will be repeated prior to each study drug administration. All patients will receive 8 cycles of oral capecitabine chemotherapy at a dose of 1250 mg/m2, administered twice daily at 12 hourly intervals for 14 consecutive days out of a 21 day cycle. Total proposed duration of therapy is 24 weeks, assuming patients commence all cycles without delay. Capecitabine and its metabolites (DFCR, DFUR and 5-FU) plasma levels will be measured during the 1st and 3rd cycles in all patients. Treatment should continue for 8 cycles unless there is evidence of disease progression, or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Surgery included proximal pancreatico-duodenectomy
* Complete macroscopic resection for ductal adenocarcinoma of the pancreas (R0 or R1 resection)
* Histological confirmation of the primary diagnosis and examination of all resection margins
* At least 4 weeks since surgery, fully recovered from the operation and fit to take part in the trial
* Age ≥ 18 years
* World Health Organisation (WHO) performance status of ≤ 2 (Appendix 1)
* Haemoglobin (Hb) ≥ 9.0 g/dl
* Neutrophils ≥ 1.5 x 109/L
* Platelets (Plts) ≥ 100 x 109/L
* Serum bilirubin ≤ 1.5 x upper normal limit
* Alanine amino-transferase (ALT) and/or aspartate amino-transferase (AST) ≤ 2.0 x upper limit of normal (ULN)
* Calculated creatinine clearance ≥ 50 ml/min (uncorrected value) or isotope clearance measurement ≥ 50ml/min
* Female patients of child-bearing potential must have a negative serum pregnancy test prior to enrolment and agree to use appropriate medically approved contraception for four weeks prior to entering the trial, during the trial and for six months afterwards.
* Male patients must agree to use appropriate medically approved contraception during the trial and for six months afterwards.
* Written, informed consent provided.
* Ability of the patient to co-operate with treatment and follow up must be ensured and documented.

Exclusion Criteria:

* Pregnancy or Lactation
* Evidence of malignant ascites, peritoneal or liver metastasis, spread to other distant abdominal or extra-abdominal organs.
* Concurrent mechanical or malabsorptive disorders precluding affective oral administration of the drug (excluding malabsorption related directly to proximal pancreatic-duodenectomy)
* Patients with pancreatic lymphoma or other histological diagnosis
* Macroscopically remaining tumour (R2 resection)
* Patients who are high medical risks because of non-malignant systemic disease including active uncontrolled infection.
* Patients with any other condition which in the Investigator's opinion would not make the patient a good candidate for the clinical trial.
* Patients known to be serologically positive for Hepatitis B, Hepatitis C or Human Immunodeficiency Virus (HIV).
* History of confirmed Ischaemic Heart Disease, concurrent congestive heart failure or prior history of class III/ IV cardiac disease (New York Heart Association [NYHA] - refer to Appendix 5)
* Any serious medical or psychological condition precluding adjuvant treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
To measure plasma levels of Capecitabine and its metabolites (DFCR, DFUR and 5-FU) | Samples collected predose and 0.25, 0.5, 1, 2, 3, 4, 5, 6, 8, and 24 hours on day 1 of cycles 1 and 3

SECONDARY OUTCOMES:
To evaluate adverse effects after every course of chemotherapy according to NCI-CTCAE V3. | 1 year (from patient registration until 28 days after last study drug administration).
To identify any dose limiting toxicities of Capecitabine | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Duncan Jodrell, DM MSc FRCP, Principal Investigator — Cambridge University Hospitals, NHS Foundation Trust, University of Cambridge
Locations (2):
- United Kingdom (2):
  - Cambridge University Hospitals NHS Foundation Trust, University of Cambridge Oncology Centre, Cambridge
  - Edinburgh Cancer Centre, Western General Hospital, Edinburgh